CLINICAL TRIAL: NCT00817986
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Tolerability of XP19986 in Subjects With Acute Back Spasms
Brief Title: A Study to Evaluate the Safety and Tolerability of Arbaclofen Placarbil (XP19986) in Subjects With Acute Back Spasms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XP-B-083
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Back Pain
Keywords: Acute back pain in the lumbar region
MeSH Terms: conditions — Back Pain | interventions — arbaclofen placarbil; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arbaclofen placarbil 20 mg (Experimental): Arbaclofen placarbil 20 mg, BID, for 14 days including the taper period.
  Interventions: Drug: Arbaclofen placarbil, 20 mg
- Placebo for Arbaclofen placarbil (Placebo Comparator): Placebo for 14 days
  Interventions: Drug: Placebo
- Arbaclofen placarbil 30 mg (Experimental): Arbaclofen placarbil 30 mg, BID, for 14 days including the taper period.
  Interventions: Drug: Arbaclofen placarbil, 30 mg
- Arbaclofen placarbil 40 mg (Experimental): Arbaclofen placarbil 40 mg, BID, for 14 days including the taper period.
  Interventions: Drug: Arbaclofen placarbil, 40 mg

INTERVENTIONS:
Drug: Arbaclofen placarbil, 20 mg — tablets
  Other Names: XP19986 SR3
  Arms: Arbaclofen placarbil 20 mg
Drug: Placebo — tablets
  Other Names: Sugar Pill
  Arms: Placebo for Arbaclofen placarbil
Drug: Arbaclofen placarbil, 30 mg — tablets
  Other Names: XP19986 SR3
  Arms: Arbaclofen placarbil 30 mg
Drug: Arbaclofen placarbil, 40 mg — tablets
  Other Names: XP19986 SR3 tablets
  Arms: Arbaclofen placarbil 40 mg

SUMMARY:
The purpose of the study is to evaluate safety and tolerability of arbaclofen placarbil sustained release tablets taken every 12 hours compared to placebo in subjects with acute back spasms in the lumbar region.

ELIGIBILITY:
Inclusion Criteria:

1. Acute moderate to severe muscle spasms in the lumbar region, as indicated by a minimum Visual Analog Scale pain severity score of 4.0 cm, beginning either:

   * within four days prior to screening for subjects who do not require a 24-hour washout

   Or
   * within three days for subjects who require a 24-hour washout
2. Willing to discontinue all analgesics (e.g. NSAIDS, COX-2 inhibitors, acetaminophen), aspirin >81 mg/day, short-acting muscle relaxants (i.e. carisoprodol, Soma®), and herbal remedies for pain at least 24 hours prior to first dose and to refrain from use during the study (cardio-protective doses of aspirin ≤ 81 mg /day are allowed).

Exclusion Criteria:

1. Clinically significant abnormal neurological history or examination at screening (excluding back spasm), including lumbar radicular symptoms, spinal stenosis, foot drop, herniated nucleus pulposus, or other structural defects
2. Subjects with back spasm related to major trauma to the region
3. Subjects with muscle spasms due to a work-related injury or subjects involved in any injury-related litigation
4. Subjects using any of the following medications at screening:

   * Opioids, both short- and long-acting including but not limited to: morphine, fentanyl patch, oxycodone, tramadol)
   * benzodiazepines, such as valium and lorazepam
   * cyclobenzaprine containing drugs (e.g., Flexeril, Amrix)
   * carisoprodol (e.g., Soma®) within 24 hours of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2008-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 14 Days
  Safety was assessed based on the incidence, intensity and relationship of treatment emergent AEs

SECONDARY OUTCOMES:
Change in pain severity score using the VAS | 4 Days

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Indivior Inc.
Locations (19):
- United States (19):
  - Litchfield Park, Arizona
  - Anaheim, California
  - San Diego, California
  - Vista, California
  - Fort Lauderdale, Florida
  - Miami, Florida
  - Atlanta, Georgia
  - Overland Park, Kansas
  - Erlanger, Kentucky
  - Traverse City, Michigan
  - Brick, New Jersey
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Oklahoma City, Oklahoma
  - Anderson, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No